CLINICAL TRIAL: NCT04000555
Title: A Randomized, Double-Blinded Placebo Controlled Study To Determine the Effectiveness of Oral Vancomycin for Secondary Prophylaxis of Clostridium Difficile Infection (CDI)
Brief Title: Oral Vancomycin for Secondary Prophylaxis of Clostridium Difficile Infection (CDI)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early due to low enrollment, this was partially related to our ability to recruit during the COVID-19 pandemic.
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00037626
Record Dates: First submitted 2019-06-17; First posted 2019-06-27 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Clostridium Difficile Infection; Clostridium Difficile Infection Recurrence
Keywords: prophylaxis
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Our primary objective is to determine the effectiveness of vancomycin in preventing recurrent Clostridium Difficile Infection (CDI) compared to placebo. Our secondary objective is to attempt to identify risk factors associated with the development of recurrent CDI.
  The purpose of this study is to gain further knowledge regarding the effectiveness of vancomycin prophylaxis in preventing Clostridium difficile infections in order to guide physicians' practices. Eligible patient's will be randomized 1:1 double-blinded placebo controlled clinical trial to determine the effectiveness of vancomycin at preventing CDI. The first arm in our study would be the "study drug" which is oral vancomycin. The second arm would be placebo. Patient with a history of CDI admitted to Tampa General Hospital or have been seen at Infectious Disease Associates of Tampa Bay clinics are receiving systemic antibiotics and have a history of at least one episode of CDI that was diagnosed on or after 4/1/2017.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators involved will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug (Experimental): Oral vancomycin 125mg twice a day prescribed for the duration of antibiotics
  Interventions: Drug: Oral Vancomycin
- Placebo (Placebo Comparator): Matched placebo twice a day prescribed for the duration of antibiotics
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Vancomycin — Oral vancomycin 125mg twice a day prescribed for the duration of antibiotics
  Arms: Study drug
Other: Placebo — Matched placebo twice a day prescribed for the duration of antibiotics
  Arms: Placebo

SUMMARY:
The purpose of this study is to gain further knowledge regarding the effectiveness of vancomycin prophylaxis in preventing Clostridium difficile infections in order to guide physicians' practices.

DETAILED DESCRIPTION:
Recurrent Clostridium difficile infection (CDI) is associated with significant morbidity, mortality and health care related costs. Up to 30% of CDI cases recur, resulting in 83,000 cases of recurrent CDI per year in the US. Although agents for primary and secondary prophylaxis for CDI including the use of probiotics, antibiotics, fecal microbiota transplantations, and newer therapies such as bezlotoxumab have been reported, there are no consensus guidelines regarding their use.

In order to understand current practices regarding secondary prophylaxis for CDI, a nationwide survey to assess physician practices regarding secondary prophylaxis for CDI. A total of 246 surveys were completed. Physicians were surveyed from greater than 100 locations. Most providers (N=173, 71%) reported using secondary prophylaxis for CDI prevention. The majority (N=138, 56%) were infectious disease providers. Vancomycin (N=121, 70%) and probiotics (N=114, 66%) were most commonly used for CDI secondary prophylaxis. Of 164 respondents who used secondary prophylaxis, 29.9% (N=49) utilized it for patients with a history of CDI who were receiving antibiotics, while 54.2% (N=89), used prophylaxis for patients with a history of recurrent CDI (more than 2 episodes) receiving antibiotics.

Despite the lack of guideline recommendations or definitive studies to support secondary prophylaxis for CDI, the majority of the physicians who responded to this survey are using secondary prophylaxis to prevent recurrent CDI. The purpose of our study is to determine the effectiveness of secondary prophylaxis with oral vancomycin vs. placebo for the prevention of recurrent clostridium difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Tampa General Hospital or outpatients at Infectious Disease Associates of Tampa Bay clinics who are receiving systemic antibiotics and have a history of at least one episode of CDI.
* Participants must at least 18 years of age to participate.
* Participants must be able to understand and sign a written informed consent form prior to initiation of study procedures.
* Expected to receive at least 3 days of systemic antibiotics.
* Life expectancy greater than 6 months.

Exclusion Criteria:

* Current CDI
* Completion of treatment for CDI within the last 15 days
* Concurrent use of drugs that have activity against C. difficile such as metronidazole, fidaxomicin, nitazoxanide, tigecycline, or rifaximine
* Concurrent use of cholestyramine
* Concurrent use of bezlotoxumab
* Concurrent use of probiotics
* Concurrent use of Imodium or other antidiarrheal agents.
* Chronic suppressive antibiotics
* Condition which causes chronic diarrhea such as inflammatory bowel disease
* Bacterial gastroenteritis other than CDI
* Pregnancy or breastfeeding
* Allergy to oral Vancomycin
* Inability to take enteric medications
* Have an unstable or life limiting condition on admission
* Already participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Recurrence Rate | 90 days
  Diagnosis of Clostridium Difficile infection to assess recurrence rates
  Participants will be called at the completion of systemic antibiotics and 1, 2 and 3 months thereafter to assess for recurrence. If participants were tested for C. difficile at another facility records will be obtained to confirm recurrent infection.

SECONDARY OUTCOMES:
Risk factors associated clostridium difficile infection recurrences | Day 0 - data will be collection upon enrollment
  Assess any risk factors associated development of recurrence such as age, number of clostridium difficile infections in the past, what antibiotics the patient has been exposed to, and exposure to proton pump inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Sampson, DO, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - Infectious Disease Associates of Tampa Bay, Tampa, Florida